CLINICAL TRIAL: NCT05593107
Title: A Study to Evaluate 68Ga-N188 PET/CT Imaging of Nectin-4 Expression in Malignant Tumors
Brief Title: 68Ga-N188 PET/CT Imaging in Malignancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jianhua ZHANG, Principal Investigator, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [68Ga]N188
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms
Keywords: [68Ga]N188; Nectin-4; PET/CT; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]N188 (Experimental): Subjects with suspected or confirmed malignancy will receive an intravenous injection of 68Ga-N188 followed by PET imaging. The subjects will also receive a whole-body 18F-FDG PET/CT scan within a one-week period.
  Interventions: Drug: [68Ga]N188

INTERVENTIONS:
Drug: [68Ga]N188 — 68Ga-N188 is injected intravenously with a dose of 0.06-0.08 mCi/kg.
  Other Names: 68Ga-N188; Nectin-4 specific PET imaging

SUMMARY:
The Nectin-4 protein belongs to the cell adhesion factors family and has a tissue-specific expression spectrum in normal human tissues. However, Nectin-4 is overexpressed in various malignancies, especially those of epithelial origins, such as uroepithelial carcinoma, making Nectin-4 a highly specific and significant imaging target for malignancies.

[68Ga]N188, a novel molecular probe of PET imaging agent that targets Nectin-4, can be used in the diagnosis and research of a wide variety of Nectin-4 high-expression malignancies, including bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed or suspected cancer;
* 18F-FDG PET/CT within 1 week;
* Signed written informed consent.

Exclusion Criteria:

* Pregnant and lactating women;
* Female patients plan to become pregnant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficacy of 68Ga-N188 PET/CT in the evaluation of malignant tumors | 1 year
  Compare the standardized Uptake Value (SUV) of lesions on 68Ga-N188 and 18F-FDG PET/CT
The diagnostic efficacy of 68Ga-N188 PET/CT in the evaluation of malignant tumors | 1 year
  Compare the number of lesions detected by 68Ga-N188 and 18F-FDG PET/CT, based on the pathology or clinical follow-up as gold standard.

SECONDARY OUTCOMES:
The dosimetry of 68Ga-N188 | 1 year
  Research on the dose distribution of 68Ga-N188 in healthy volunteers and cancer patients by 1-hour dynamic PET/CT acquisition and analyze by the dosimetry software
Quantitative evaluation of 68Ga-N188 | 1 year
  Evaluation of quantitative parameters of 68Ga-N188, such as time-activity curve.
Correlation with pathological expression | 1 year
  Analyze Nectin-4 expression at the imaging level in combination with Nectin-4 expression in pathological specimens

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China